CLINICAL TRIAL: NCT06612060
Title: Comparative Randomized Study of Blood Coagulation Triggering and Thromboresistance of Biocompatible Versus Non-coated Extracorporeal Circuits During Cardiac Surgery
Brief Title: Biocompatible Versus Non-coated Extracorporeal Circuits in Cardiac Surgery
Acronym: BALANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polychronis Antonitsis (Other)
Responsible Party: Sponsor-Investigator, Polychronis Antonitsis, Associate Professor of Cardiac Surgery, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BALANCE_CTS
Record Dates: First submitted 2024-09-09; First posted 2024-09-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery Requiring Cardiopulmonary Bypass; Extracorporeal Circulation
Keywords: Bio-compatible; Surface Coating; Thromboresistance; Coagulation; cardiopulmonary bypass; extracorporeal circulation; cardiac surgery
MeSH Terms: conditions — Thrombosis | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coated circuit (Experimental): Cardiac surgery with a specialized biocompatible extracorporeal circulation circuit with a hydrophobic coating.
  Interventions: Procedure: Cardiac surgery with the use of extracorporeal circulation
- Non-coated circuit (Active Comparator): Cardiac surgery with the conventional non-coated extracorporeal circulation circuit.
  Interventions: Procedure: Cardiac surgery with the use of extracorporeal circulation

INTERVENTIONS:
Procedure: Cardiac surgery with the use of extracorporeal circulation — All randomized patients will undergo open heart surgery with the use of extracorporeal circulation. Criteria for randomization: i) age between 18 and 80 years and ii) elective procedure.

SUMMARY:
The aim of the present strudy is to investigate whether the use of biocompatible extracorporeal circulation circuits with a special hydrophilic polymer coating without heparin causes a reduction in the activation of the coagulation mechanism and the formation of microthrombi in the circuit tubing. A total of 50 patients undergoing cardiac surgery with extracorporeal circulation will be randomized in two groups using a computer-generated algorithm. The first group (study group) will undergo cardiac surgery with a specialized biocompatible circuit with a hydrophilic coating, while the control group will be operated with the conventional non-coated extracorporeal circulation circuit. During the period of extracorporeal circulation, blood samples will be taken at predetermined times which will be analyzed with the ELISA technique to determine the levels of prothrombin fragments 1+2 (F1+2), thrombin/antithrombin complex (TAT) as well as platelet factor P-selectin. Moreover, sections of the circuit tubes will be examined under electron microscopy for quantitative evaluation of microthrombi detected on the walls. The expected outcome of the study is to establish, with the use of specific biochemical markers and electron microscopy the protective effect of biocompatible coated extracorporeal circulation circuits on the coagulation mechanism and platelet activation.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgery

Exclusion Criteria:

* Need for emergency surgery
* Serious hematological condition causing anemia, thrombocytopenia, etc.
* Receiving immunosuppressive treatment
* Inability to obtain consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prothrombin fragments 1+2 (F1+2) | Change from baseline at 40 and 80 minutess after initiation of extracorporeal circulation
  Plasma levels of prothrombin fragments 1+2 (F1+2) (pg/ml) will be calculated at predetermined times using the ELISA technique
Thrombin/Antithrombin complex (TAT) | Change from baseline at 40 and 80 minutess after initiation of extracorporeal circulation
  Plasma levels of thrombin/antithrombin complex (TAT) (pg/ml) will be calculated at predetermined times using the ELISA technique
Platelet factor P-selectin | Change from baseline at 40 and 80 minutes after initiation of extracorporeal circulation
  Plasma levels of platelet factor P-selectin (pg/ml) will be calculated at predetermined times using the ELISA technique
Circuit microthrombi | Immediately after the cessation of cardiopulmonary bypass.
  Quantitative evaluation of microthrombi on the walls of the circuit tubes as detected by electron microscopy.

SECONDARY OUTCOMES:
Mortality | From the day of surgery up to 30 postoperative days
  Death from any cause
Transfusion | From the day of surgery until the day of discharge from hospital, assessed up to one month.
  Incidence of blood product (RBC, FFP, platelet) transfusion
Major morbidity | From the day of surgery until the day of discharge from hospital, assessed up to one month.
  Composite outcome consisting of: stroke, myocardial infarction, need for revascularization, acute renal failure, prolonged > 48 h need for mechanical ventilation, reoperation).
Bleeding | 12 hours after surgery
  Volume of blood collected at the chest tubes.
ICU stay | From the day of surgery until the day of discharge from hospital, assessed up to one month.
  ICU stay in hours.
Hospital stay | From the day of surgery until the day of discharge from hospital, assessed up to one month.
  Total hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Isaak Keremidis, MScP, Principal Investigator — Aristotle University Of Thessaloniki; Polychronis Antonitsis, MD, PhD, Study Chair — Aristotle University of Theesaloniki School of Medicine; Kali Makedou, MD, PhD, Study Director — Aristole University of Thessaloniki School of Medicine; Theodora Papamitsou, MD, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- Interbalkan Hospital, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gore S, Andersson J, Biran R, Underwood C, Riesenfeld J. Heparin surfaces: Impact of immobilization chemistry on hemocompatibility and protein adsorption. J Biomed Mater Res B Appl Biomater. 2014 Nov;102(8):1817-24. doi: 10.1002/jbm.b.33154. Epub 2014 Apr 8. PMID 24711209
- [Background] Modrau IS, Halle DR, Nielsen PH, Kimose HH, Greisen JR, Kremke M, Hvas AM. Impact of minimally invasive extracorporeal circulation on coagulation-a randomized trial. Eur J Cardiothorac Surg. 2020 Jun 1;57(6):1145-1153. doi: 10.1093/ejcts/ezaa010. PMID 32011717
- [Background] Teligui L, Dalmayrac E, Mabilleau G, Macchi L, Godon A, Corbeau JJ, Denomme AS, Bouquet E, Boer C, Baufreton C. An ex vivo evaluation of blood coagulation and thromboresistance of two extracorporeal circuit coatings with reduced and full heparin dose. Interact Cardiovasc Thorac Surg. 2014 Jun;18(6):763-9. doi: 10.1093/icvts/ivu011. Epub 2014 Mar 14. PMID 24632424